CLINICAL TRIAL: NCT05349968
Title: A Clinical Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Multiple Dosing of Lipovirtide for Injection in HIV-infected Patients Who Have Not Received Antiretroviral Therapy
Brief Title: Pharmacokinetics and Efficacy of Multiple Dosing of Lipovirtide for Injection in HIV-infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanxi Kangbao Biological Product Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB-LP-80-102
Record Dates: First submitted 2022-04-02; First posted 2022-04-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose 5 mg (Experimental): Injected subcutaneously at room temperature into the abdomen (moles, scar tissue, bruises or areas other than the navel) and administered once a week for 4 weeks, with no more than 2.0 mL volume administered to a single site.
  Interventions: Drug: Lipovirtide for injection
- Dose 20 mg (Experimental): Injected subcutaneously at room temperature into the abdomen (moles, scar tissue, bruises or areas other than the navel) and administered once a week for 4 weeks, with no more than 2.0 mL volume administered to a single site.
  Interventions: Drug: Lipovirtide for injection
- Dose 40 mg (Experimental): Injected subcutaneously at room temperature into the abdomen (moles, scar tissue, bruises or areas other than the navel) and administered once a week for 4 weeks, with no more than 2.0 mL volume administered to a single site.
  Interventions: Drug: Lipovirtide for injection

INTERVENTIONS:
Drug: Lipovirtide for injection — Multiple dosing of Lipovirtide
  Other Names: nothing

SUMMARY:
Primary Objectives

1.Evaluation of safety and tolerability after repeated administration of injectable Lipivirtide in HIV-infected patients not receiving antiretroviral therapy

Secondary Objectives

1. Evaluation of the pharmacokinetic properties of injectable Lipovirtide after multiple administrations in HIV-infected patients not receiving antiretroviral therapy, to obtain pharmacokinetic parameters.
2. Evaluation of the efficacy of injectable Lipovirtide for HIV in HIV-infected patients not receiving antiretroviral therapy.
3. Evaluation of the immunogenicity of lipovirtide for injection.

DETAILED DESCRIPTION:
PK parameters were calculated by Phoenix WinNonlin 8.2 (or higher) and other data were analyzed using SAS 9.4 (or higher) software.

Full analysis set: will be used for efficacy analysis. Descriptive statistics of HIV viral load and CD4+ T-cell count at each time point, calculation of subject means, standard deviations, quartiles, minimum and maximum values, and comparison of changes from baseline at each time point.

Safety analysis set: calculation of the incidence of adverse events and systematic categorization. Calculate the incidence of adverse events and systematically categorize them. Cross tabulation of clinical determination before and after drug administration for laboratory tests, ECG tests, and physical examination. Changes in measured values of vital signs over time. The actual measured values of the vital signs varied over time.

Immunogenicity analysis: statistics of the results of each indicators (including the positive incidence and titer) over time, and a detailed list of the results of each visit.

Pharmacokinetic analysis: individual and mean c-t curves were plotted; mean, standard deviation, interquartile, maximum, minimum and coefficient of variation of blood concentrations at each time point were listed. Pharmacokinetic parameters were calculated for each subject from the non-compartment model. and the arithmetic mean, standard deviation, quartiles, maximum value, minimum value and geometric mean and coefficient of variation were also calculated for each parameter.

ELIGIBILITY:
Inclusion Criteria:

1. 18~60 years old (including the critical value), male and female are not limited.
2. Body mass index BMI [weight (kg)/height2 (m2)] is 18.0~28.0 (including the critical value), male weight should be ≥50kg, female weight should be ≥45kg.
3. Diagnosed with HIV-1 infection.
4. Those who did not plan to have children within 2 weeks prior to screening and within 3 months after the end of the trial and who agreed to use effective non-pharmacological contraception during the trial.
5. Subjects should fully understand the purpose, nature and methods of the test and the possible adverse effects and voluntarily participate in this test.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be allowed to enter the trial

1. The presence of any of the following 1）Unexplained persistent irregular fever of 38°C or more for >1 month. 2）Diarrhea (stools more than 3 times/day), >1 month. 3）Weight loss of 10% or more within 6 months. 4）Recurrent oral fungal infections. 5）Recurrent herpes simplex virus infection or herpes zoster virus infection. 6）Pneumocystis carinii pneumonia (PCP). 7）Recurrent bacterial pneumonia. 8）Active tuberculosis or non-tuberculous mycobacteriosis. 9）Deep fungal infection. 10）Occupational lesions of the central nervous system. 11）Dementia in young and middle-aged adults. 12）Active cytomegalovirus (CMV) infection. 13）Toxoplasma encephalopathy. 14）Malnefield basket disease. 15）Recurrent sepsis. 16）Kaposi's sarcoma, lymphoma.
2. Patients who have received antiviral therapy and/or HIV vaccination;
3. HBsAg of (+), and/or anti-HCV of (+);
4. Abnormal liver function (ALT/AST>3XULN, or TBIL>2XULN);
5. Creatinine clearance<70mL/min (Equation of calculation: Cockcroft-Gault)
6. Existing severe chronic disease, metabolic disease (such as diabetes), neurological and psychiatric disease;
7. History of pancreatitis;
8. Regnant, lactating women and women of childbearing age who cannot use contraception as required;
9. People with allergies or known allergies to the ingredients of this medicine;
10. People with a history of smoking within 12 months before screening (the average number of cigarettes smoked per day is 35.);
11. People with a history of alcoholism within 12 months before screening(Drink N14 units of alcohol per week on average: 1 unit = 285mL of beer, or 25mL of spirits, or 150mL of wine) or positive alcohol breath test before enrollment;
12. People with have a history of drug abuse within 12 months before screening or those who tested positive for addictive substances before enrollment;
13. Participated in other drug trials within 3 months before screening;
14. The investigator believes that the subject has other conditions that are not suitable for participating in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in respiration rate of Vital Signs. | Within 50 days after the first administration.
  Respiration rate in times / minute
Changes from baseline in Blood lactate of Laboratory Examination. | Within 50 days after the first administration.
  Changes of blood lactate will be recorded.
Changes from baseline in Pregnancy test of Laboratory Examination. | Within 50 days after the first administration.
  Pregnancy test will be tested in female subjects.
Changes from baseline in Drug resistance test of Laboratory Examination. | Within 50 days after the first administration.
  Changes of drug resistance test will be recorded.Evaluate the proportion of HIV resistance in subjects.
Changes from baseline in Immunogenic blood collection of Laboratory Examination. | Within 50 days after the first administration.
  Changes of immunogenic blood collection will be recorded.The historical changes of test results (including positive rate and titer) of various indicators were counted.
Changes from baseline in blood pressure of Vital Signs. | Within 50 days after the first administration.
  Blood pressure in mmHg
Changes from baseline in body temperature of Vital Signs. | Within 50 days after the first administration.
  Body temperature in Celsius degree
Changes from baseline in red blood cell count of Laboratory Examination. | Within 50 days after the first administration.
  Red blood cell count in whole blood is reported in the form of number.
Changes from baseline in white blood cell count of Laboratory Examination. | Within 50 days after the first administration.
  White blood cell count in whole blood is reported in the form of number.
Changes from baseline in neutrophil count of Laboratory Examination. | Within 50 days after the first administration.
  Neutrophil count in whole blood is reported in the form of number.
Changes from baseline in lymphocyte count of Laboratory Examination. | Within 50 days after the first administration.
  Lymphocyte count in whole blood is reported in the form of number.
Changes from baseline in platelet count of Laboratory Examination. | Within 50 days after the first administration.
  Platelet count in whole blood is reported in the form of number.
Changes from baseline in hemoglobin of Laboratory Examination. | Within 50 days after the first administration.
  Changes of hemoglobin concentration（g/dL）in whole blood will be recorded.
Changes from baseline in PT of Laboratory Examination. | Within 50 days after the first administration.
  Prothrombin time (PT) is a screening test for exogenous coagulation factors.
Changes from baseline in INR of Laboratory Examination. | Within 50 days after the first administration.
  International standardized ratio (INR) is calculated from prothrombin time and international sensitivity index (ISI) of the reagent.
Changes from baseline in APTT of Laboratory Examination. | Within 50 days after the first administration.
  Activated partial thromboplastin time (APTT) is a screening test for endogenous coagulation factors.
Changes from baseline in total bilirubin of Laboratory Examination. | Within 50 days after the first administration.
  Changes of total bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in direct bilirubin of Laboratory Examination. | Within 50 days after the first administration.
  Changes of direct bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in ALT of Laboratory Examination. | Within 50 days after the first administration.
  Changes of ALT concentration (U/L) in serum will be recorded.
Changes from baseline in AST of Laboratory Examination. | Within 50 days after the first administration.
  Changes of AST concentration (U/L) in serum will be recorded.
Changes from baseline in total protein of Laboratory Examination. | Within 50 days after the first administration.
  Changes of total protein concentration (g/L) in serum will be recorded.
Changes from baseline in albumin of Laboratory Examination. | Within 50 days after the first administration.
  Changes of albumin concentration (g/L) in serum will be recorded.
Changes from baseline in total bile acid of Laboratory Examination | Within 50 days after the first administration.
  Changes of total bile acid concentration (μmol/L) in serum will be recorded.
Changes from baseline in urea of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urea concentration (mmol/L) in serum will be recorded.
Changes from baseline in creatinine of Laboratory Examination. | Within 50 days after the first administration.
  Changes of creatinine concentration (μmol/L) in serum will be recorded.
Changes from baseline in uric acid of Laboratory Examination. | Within 50 days after the first administration.
  Changes of uric acid concentration (μmol/L) in serum will be recorded.
Changes from baseline in glucose of Laboratory Examination | Within 50 days after the first administration.
  Changes of glucose concentration (mmol/L) in serum will be recorded.
Changes from baseline in potassium of Laboratory Examination. | Within 50 days after the first administration.
  Changes of potassium concentration (mmol/L) in serum will be recorded.
Changes from baseline in sodium of Laboratory Examination. | Within 50 days after the first administration.
  Changes of sodium concentration (mmol/L) in serum will be recorded.
Changes from baseline in chlorine of Laboratory Examination. | Within 50 days after the first administration.
  Changes of chlorine concentration (mmol/L) in serum will be recorded.
Changes from baseline in urine specific gravity of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urine specific gravity will be recorded.
Changes from baseline in urine pH of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urine pH value will be recorded.
Changes from baseline in urine glucose of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urine glucose will be examined by qualitative test (positive or negative).
Changes from baseline in urine protein of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urine protein will be examined by qualitative test (positive or negative).
Changes from baseline in urine ketone body of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urine ketone body will be examined by qualitative test (positive or negative).
Changes from baseline in urine white blood cell of Laboratory Examination. | Within 50 days after the first administration.
  Changes of white blood cell in urine will be examined by qualitative test (positive or negative).
Changes from baseline in urine bilirubin of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urine bilirubin will be examined by qualitative test (positive or negative).
Changes from baseline in urine occult blood of Laboratory Examination. | Within 50 days after the first administration.
  Changes of urine occult blood will be examined by qualitative test (positive or negative).
Changes from baseline in Electrocardiogram. | Within 50 days after the first administration.
  The cardiac rhythm is showed in electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded，To evaluate the incidence of abnormal electrocardiogram.
Changes from baseline in CK of Laboratory Examination | Within 50 days after the first administration.
  Changes of CK concentration (U/L) in serum will be recorded.
Changes from baseline in CK-MB of Laboratory Examination | Within 50 days after the first administration.
  Changes of CK-MB concentration (ng/mL) in serum will be recorded.
Changes from baseline in LDH of Laboratory Examination | Within 50 days after the first administration.
  Changes of LDH concentration (U/L) in serum will be recorded.
Changes from baseline in ALP of Laboratory Examination | Within 50 days after the first administration.
  Changes of ALP concentration (U/L) in serum will be recorded.
Changes from baseline in Triglyceride of Laboratory Examination | Within 50 days after the first administration.
  Changes of Triglyceride concentration (mmol/L) in serum will be recorded.
Changes from baseline in CHOL of Laboratory Examination | Within 50 days after the first administration.
  Changes of CHOL concentration (mmol/L) in serum will be recorded.
Changes from baseline in TP of Laboratory Examination | Within 50 days after the first administration.
  Changes of TP concentration (g/L) in serum will be recorded.
Changes from baseline in ALB of Laboratory Examination | Within 50 days after the first administration.
  Changes of ALB concentration (g/L) in serum will be recorded.
Changes from baseline in UA of Laboratory Examination | Within 50 days after the first administration.
  Changes of UA concentration (μmol/L) in serum will be recorded.
Changes from baseline in GLU of Laboratory Examination | Within 50 days after the first administration.
  Changes of GLU concentration (mmol/L) in serum will be recorded.
Changes from baseline in AMY of Laboratory Examination | Within 50 days after the first administration.
  Changes of AMY concentration (U/L) in serum will be recorded.

SECONDARY OUTCOMES:
Changes from baseline in HIV viral load detection of Laboratory Examination. | Within 50 days after the first administration.
  Changes of HIV viral load detection will be recorded.
Changes from baseline in CD4+T cell counts of Laboratory Examination. | Within 50 days after the first administration.
  Changes of CD4+T cell counts will be recorded.
Incidence of anti-Lipovetin antibody. | Within 50 days after the first administration.
  Incidence of anti-Lipovetin antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Yu, Principal Investigator — Beijing You'an Hospital, Beijing Medical University; Hao Wu, Principal Investigator — Beijing You'an Hospital, Beijing Medical University
Locations (1):
- Beijing You'an Hospital, Beijing Medical University, Beijing, China